CLINICAL TRIAL: NCT07175844
Title: Comparative Effects of Vocal and Breathing Exercises on Respiratory Function and Trunk Stability in Women
Acronym: VO vs BE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: LithuanianSportsU-25
Record Dates: First submitted 2025-09-02; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Healthy Subjects
Keywords: women; vocal exercises; breathing exercises; core stability; spirometry
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VE group (Experimental): Participants performed six weekly sessions of 30 minutes, guided by videos focusing on diaphragmatic breathing and contemporary singing techniques. Initial exercises (weeks 1-2) included sustained "s" sounds, lip trills, humming, melodic vowel sequences, and "Ja" exercises. Weeks 3-6 included advanced solo exercises such as short and long "S", humming variations, "mum" vocalizations, rhythmic patterns ("cha-cha-cha"), melodic sequences ("Niemak 1-3"), and counting exercises. Exercises were performed standing, preferably in front of a mirror.
  Interventions: Other: Vocal exercises
- BE group (Active Comparator): Participants in the breathing exercises group were given access to a 30-minute instructional video, in which a licensed physiotherapist demonstrated how to perform the exercises. Participants were instructed to complete the exercises twice per week at a time convenient for them. They could reflect on the exercises and submit questions to the physiotherapist within a closed social media group. Two weeks after the start of the intervention, participants were advised to increase the intensity of the exercises: lengthening inhalation, exhalation, and breath-holding during square breathing, and increasing the number of exhalations during "Kapalabhati" breathing from 20 to 60 per series, while respecting individual comfort and tolerance.
  Interventions: Other: Breathing exercises

INTERVENTIONS:
Other: Vocal exercises — Participants performed six weekly sessions of 30 minutes, guided by videos focusing on diaphragmatic breathing and contemporary singing techniques. Initial exercises (weeks 1-2) included sustained "s" sounds, lip trills, humming, melodic vowel sequences, and "Ja" exercises. Weeks 3-6 included advanced solo exercises such as short and long "S", humming variations, "mum" vocalizations, rhythmic patterns ("cha-cha-cha"), melodic sequences ("Niemak 1-3"), and counting exercises. Exercises were performed standing, preferably in front of a mirror.
  Arms: VE group
Other: Breathing exercises — Participants in the breathing exercises group were given access to a 30-minute instructional video, in which a licensed physiotherapist demonstrated how to perform the exercises. Participants were instructed to complete the exercises twice per week at a time convenient for them. They could reflect on the exercises and submit questions to the physiotherapist within a closed social media group. Two weeks after the start of the intervention, participants were advised to increase the intensity of the exercises: lengthening inhalation, exhalation, and breath-holding during square breathing, and increasing the number of exhalations during "Kapalabhati" breathing from 20 to 60 per series, while respecting individual comfort and tolerance.
  Arms: BE group

SUMMARY:
The goal of this randomized clinical trial is to investigate whether vocal exercises or breathing exercises improve respiratory function and trunk stability in healthy adult women aged 18-65. The main questions it aims to answer are:

Do vocal exercises improve respiratory function, respiratory muscle strength, endurance, and trunk stability? Do breathing exercises improve respiratory function, respiratory muscle strength, and endurance? Researchers will compare the vocal exercises group to the breathing exercises group to determine if one intervention has a superior effect on lung function, respiratory muscle performance, and trunk stability.

Participants will:

Perform a 6-week program of either vocal exercises or breathing exercises, with sessions twice per week, 30 minutes each.

Complete pre- and post-intervention assessments including thoracic excursion, breath-hold tests, spirometry, Dynamic Neuromuscular Stabilization (DNS) tests, and trunk stability tests using the Stabilizer pressure biofeedback device.

Engage with instructional videos and guidance through a closed social media group, allowing questions and feedback to ensure correct technique.

DETAILED DESCRIPTION:
Study Design This study was a randomized controlled trial designed to evaluate the effects of vocal exercises versus breathing exercises on respiratory function and trunk stability in adult women. Ethical approval was obtained from the [name of ethics committee] (Approval No.: 2024 12 09 MNL-KIN (M)-2024-726). All participants provided written informed consent prior to enrollment, in accordance with the Declaration of Helsinki.

Participants Fifty healthy women aged 18-65 years were recruited via an online questionnaire distributed on social media. Inclusion criteria were female sex, age 18-65 years, no prior engagement in structured breathing or vocal training in the previous six months, and absence of acute or chronic respiratory infection. Exclusion criteria included inability to attend in-person assessments or failure to meet age or health criteria. Baseline demographic characteristics (age, weight, height, BMI) were comparable between groups.

Randomization and Allocation Eligible participants (n = 50) were randomly assigned in a 1:1 ratio to either the Vocal Exercises Group (VE, n = 25) or the Breathing Exercises Group (BE, n = 25) using a computer-generated random sequence. Both interventions lasted six weeks, with participants completing sessions twice per week for 30 minutes each.

Intervention

Breathing Exercises Group

Participants were provided access to a 30-minute instructional video demonstrating the following exercises:

Conscious Breathing: Seated observation of chest and abdominal wall movement.

Humming Bee (Bhramari Pranayama): Exhalation with a humming sound and ears gently occluded.

Kapalabhati: Rapid forceful exhalations with passive inhalations; intensity increased over time.

Alternate Nostril Breathing (Nadi Shodhana): Cycles of inhalation and exhalation through alternate nostrils.

Square Breathing (4x4x4x4): Seated breathing with equal durations of inhalation, breath-hold, exhalation, and breath-hold.

Diaphragmatic Breathing: Supine breathing with lateral rib expansion.

Vocal Exercises Group

Participants received access to instructional videos emphasizing diaphragmatic breathing and contemporary singing techniques. Exercises included:

Initial Exercises (Weeks 1-2): Sustained "s" sounds, lip trills, humming, melodic vowel sequences, and short vocal phrases.

Solo Vocal Exercises (Weeks 3-6): Short and long "S" sounds, humming on single and multiple notes, "mum" vocalization sequences, "Cha-cha-cha" sequences, melodic humming, and counting exercises without inhalation.

Both groups had access to a closed social media group for guidance and questions. Intensity adjustments were recommended after two weeks based on participant tolerance.

Outcome Measures Assessments were conducted at baseline and after six weeks.

Respiratory Function

Thoracic Excursion (CE): Measured at Th3-4, Th7-8, and Th11-12 using a tape measure. CE was calculated as the difference between maximal inspiration and expiration.

Spirometry: FEV₁, FVC, and PEF were measured using a handheld wireless spirometer (Contec SP80B). Three trials were performed, and the mean value was used.

Breath-Hold Tests: Stange (after maximal inspiration) and Genchi (after maximal expiration) tests were conducted in a seated position.

Trunk Stability

Dynamic Neuromuscular Stabilization (DNS): Three tests were used-diaphragm function, head/neck/trunk flexion, and head/neck/trunk extension. Tests were scored on a 4-point scale (1 = failed, 4 = excellent).

Stabilizer Pressure Biofeedback Device: Four tests assessed trunk stability: prone, supine, bent-leg lift, and straight-leg lift. Mean pressure differences over three repetitions were calculated for each leg.

Statistical Analysis Data were analyzed using IBM SPSS Statistics 29.0. Normality was confirmed using the Shapiro-Wilk test (p > 0.05). Within-group comparisons were performed with paired-samples t-tests, and between-group differences were assessed using independent-samples t-tests. Statistical significance was set at p < 0.05. Effect sizes were interpreted according to Cohen's d: 0.00-0.20 = no effect, 0.21-0.50 = small, 0.51-0.80 = medium, 0.81-1.30 = large, >1.30 = very large.

Flow of Participants Eighty-six participants were initially screened; 26 were excluded (19 due to recent training, 6 unable to attend in-person, 1 outside age range). Fifty participants were randomized and completed the six-week intervention with no attrition.

ELIGIBILITY:
Inclusion Criteria:

* female sex;
* age 18-65 years;
* no engagement in breathing exercises for at least six months;
* no engagement in vocal training for at least six months;

Exclusion Criteria:

* acute respiratory diseases.
* chronic respiratory diseases

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume (FEV₁) | 6 weeks
  Forced expiratory volume (FEV₁) was measured in liters in one second (L/s) using the Contec Spirometer SP80B. Three trials were performed per participant, with the mean used for analysis.
Stange test | 6 weeks
  The Stange test (breath-hold after maximal inhalation) was performed in a seated position. Before testing, participants were instructed to breathe calmly, and breath-hold duration (in seconds) was recorded using a stopwatch.
Forced vital capacity (FVC) | 6 weeks
  Forced vital capacity (FVC) was measured in liters (L) with Contec Spirometer SP80B. Three trials were performed per participant, with the mean used for analysis.
Peak expiratory flow (PEF) | 6 weeks
  Peak expiratory flow (PEF) was measured in liters per one second (L/s) using the Contec Spirometer SP80B. Three trials were performed per participant, with the mean used for analysis.
Genchi test | 6 weeks
  The Genchi test (breath-hold after maximal exhalation) waas performed in a seated position. Before testing, participants were instructed to breathe calmly, and breath-hold duration (in seconds) was recorded using a stopwatch.

SECONDARY OUTCOMES:
Dynamic Neuromuscular Stabilization (DNS) | 6 weeks
  Three DNS functional tests were selected: the diaphragm test, head/neck/trunk flexion test, and head/neck/trunk extension test (Kobesova et al., 2020). Tests were scored on a 4-point scale (1 = failed, 4 = excellent) based on muscle activation, symmetry, posture, and compensatory movements.
Trunk Stability Tests | 6 weeks
  Trunk stability was assessed using the Stabilizer Pressure Bio-Feedback device. Four tests were conducted: prone activation, supine activation, bent-leg lift, and straight-leg lift. Pressure changes during abdominal muscle activation were recorded, with three repetitions per test and mean values calculated (Garnier, 2009; Herrington, 2005).

CONTACTS AND LOCATIONS:
Overall Officials: Eirida S Kudirkienė, MSc, Principal Investigator — Lithuanian Sports University
Locations (2):
- Lithuania (2):
  - Department of Health Promotion and Rehabilitation, Kaunas, Lithuania
  - Lithuanian Sports University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided